CLINICAL TRIAL: NCT04727554
Title: A Phase 1, Multicenter, Open-label, Dose Exploration and Dose Expansion Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of AMG 994 Monotherapy and Combination of AMG 994 and AMG 404 in Subjects With Advanced Solid Tumors
Brief Title: Study of AMG 994 Monotherapy and AMG 994 and AMG 404 Combination Therapy in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20190136
Record Dates: First submitted 2021-01-25; First posted 2021-01-27 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumors
Keywords: Mesothelin expression

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1a: Dose Exploration (Experimental): Determine the maximum tolerated dose (MTD) or the recommended phase 2 dose (RP2D) of AMG 994, in combination with AMG 404.
  Interventions: Drug: AMG 994; Drug: AMG 404
- Part 1b: Dose Exploration (Experimental): Determine the maximum tolerated dose (MTD) or the recommended phase 2 dose (RP2D) of AMG 994, in combination with AMG 404.
  Interventions: Drug: AMG 994; Drug: AMG 404
- Part 1c: Dose Exploration (Experimental): Determine the maximum tolerated dose (MTD) or the recommended phase 2 dose (RP2D) of AMG 994, in combination with AMG 404.
  Interventions: Drug: AMG 994; Drug: AMG 404
- Part 2: Dose Expansion (Experimental): Participants will be administered with the MTD or RP2D of AMG 994 identified in the dose escalation part of the study, in combination with AMG 404.
  Interventions: Drug: AMG 994; Drug: AMG 404

INTERVENTIONS:
Drug: AMG 994 — Administered as an intravenous (IV) infusion.
Drug: AMG 404 — Administered as an intravenous (IV) infusion.

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability, and maximum tolerated dose (MTD)/maximum tolerated combination dose (MTCD) or recommended phase 2 dose (RP2D) of AMG 994 as monotherapy and AMG 994 in combination with AMG 404 in participants with advanced solid tumors.

DETAILED DESCRIPTION:
AMG 994 will be administered by short term intravenous (IV) infusion once weekly in each 28-day cycle and AMG 404 will be administered by short-term IV infusion once every 4 weeks (Q4W) in a 28 day cycle (on day 1 of cycle 2 and beyond). The study will be conducted in 2 parts: Part 1 - Dose Exploration and Part 2 - Dose Expansion.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent/assent prior to initiation of any study specific activities/procedures.
* Age ≥ 18 years at the time of signing informed consent.
* Life expectancy of > 3 months, in the opinion of the investigator.
* Participant must have histologically or cytologically proven metastatic or locally advanced solid tumors of known MSLN expression who have relapsed after and/or are refractory to established and available therapies with known clinical benefit, for which:

  * No standard systemic therapy exists; or
  * Standard systemic therapy has failed or is not available.
* Dose Expansion (Part 2): Participant must have one of the following malignancies: mesothelioma, pancreatic adenocarcinoma, MSLN positive NSCLC squamous cell carcinoma or adenocarcinoma, high grade serous ovarian carcinoma.
* At least 1 measurable or evaluable lesion as defined by modified RECIST 1.1 guidelines.
* Participants must be willing to undergo a biopsy prior to enrollment and during treatment with AMG 994.
* Participants with treated brain metastases are eligible provided they meet the following criteria:

  * Definitive therapy was completed at least 2 weeks prior to enrollment.
  * No evidence of radiographic central nervous system (CNS) progression or CNS disease following definitive therapy and by the time of study screening. Patients manifesting progression in lesions previously treated with stereotactic radiosurgery may still be eligible if pseudoprogression can be demonstrated by appropriate means and after discussion with the medical monitor.
  * Any CNS disease is asymptomatic, any neurologic symptoms due to CNS disease have returned to baseline, or non-serious CNS diseases that are asymptomatic and deemed irreversible (eg, peripheral neuropathy), the patient is off steroids for at least 7 days (physiologic doses of steroids are permitted), and the patient is off or on stable doses of anti-epileptic drugs for malignant CNS disease and has not had a seizure within 1 month prior to the screening visit.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
* Hematologic function, as follows (transfusions or growth factor support must not be administered within 7 days prior to obtaining screening labs):

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 75 x 109/L
  * Hemoglobin ≥ 9 g/dL
* Adequate renal laboratory assessments, as follows:

  • Estimated glomerular filtration rate based on Modification of Diet in Renal Disease (MDRD) calculation ≥ 45 mL/min/1.73 m2
* Hepatic function, as follows:

  * Total bilirubin (TBL) ≤ 1.5 x upper limit of normal (ULN) or ≤ 3 x ULN for participants with liver metastasis
  * Aspartate transaminase (AST) ≤ 3 x ULN or ≤ 5 x ULN for participants with liver metastasis
  * Alanine aminotransferase (ALT) ≤ 3 x ULN or ≤ 5 x ULN for participants with liver metastasis
  * Alkaline phosphatase ≤ 2.5 x ULN or ≤ 5 x ULN for participants with liver metastasis

Exclusion Criteria:

Disease Related

* Primary brain tumor, untreated or symptomatic brain metastases and leptomeningeal disease.

Other Medical Conditions

* History of other malignancy within the past 2 years, with the following exception[s]:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before enrollment and felt to be at low risk for recurrence by the treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated cervical carcinoma in situ without evidence of disease.
  * Adequately treated breast ductal carcinoma in situ without evidence of disease.
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer.
  * Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ.
* Participants with NSCLC squamous cell carcinoma (Part 1), MSLN negative NSCLC squamous cell carcinoma (Part 2), or MSLN negative NSCLC adenocarcinoma (Part 2) once the participant has been screened for MSLN expression.
* Participants with sarcomatoid mesothelioma and small cell lung cancer will be excluded from both the Dose Exploration (Part 1) and Dose Expansion (Part 2) parts of the study.
* History of solid organ transplantation.
* Major surgery within 28 days of study day 1.

Prior/Concomitant Therapy

* Anti-tumor therapy (radiotherapy, chemotherapy, antibody therapy, molecular targeted therapy, or investigational agent) within 21 days prior to study day 1.
* Treatment with a checkpoint inhibitor within 9 weeks prior to study day 1.
* Live vaccine therapy within 4 weeks prior to study drug administration.
* Current treatment or within 14 days of day 1 with immunosuppressive corticosteroid defined as > 10 mg prednisone daily or equivalent. Steroids with no minimal systemic effect (such as topical or inhalation) are permitted.

Prior/Concurrent Clinical Study Experience

* Currently receiving treatment in another investigational device or drug study, or less than 21 days prior to study day 1 since ending treatment on another investigational device or drug study(ies).
* Evidence of active or radiological sequelae of non-infectious pneumonitis.
* History of any immune-related colitis. Infectious colitis is allowed if evidence of adequate treatment and clinical recovery exists and at least 3 months interval observed since diagnosis of colitis.
* History of allergic reactions or acute hypersensitivity reaction to antibody therapies.
* Positive/non-negative test results for human immunodeficiency virus (HIV).
* Hepatitis B and C based on the following results:

  * Positive for hepatitis B surface antigen (HBsAg) (indicative of chronic hepatitis B or recent acute hepatitis B)
  * Negative HBsAG and positive for hepatitis B core antibody: hepatitis B virus DNA by polymerase chain reaction (PCR) is necessary. Detectable hepatitis B virus DNA suggests occult hepatitis B.
  * Positive hepatitis C virus antibody (HCVAb): hepatitis C virus RNA by PCR is necessary. Detectable hepatitis C virus RNA suggests chronic hepatitis C.
* Active infection requiring oral or intravenous therapy.
* Active or history of any autoimmune disease or immunodeficiencies. Participants with diabetes Type 1, vitiligo, psoriasis, hypo- or hyper-thyroid disease not requiring immunosuppressive treatment are permitted.
* Myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or cardiac arrhythmia requiring medication.
* Unresolved toxicities from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 1, or are stable and well controlled with minimal, local, or noninvasive intervention AND there is agreement to allow by both the investigator and the Amgen Medical Monitor.

  * Any history of grade 3 or higher colitis, pneumonitis, or neurological toxicity OR
  * Unresolved toxicities from prior checkpoint inhibitor therapy, defined as not having resolved to CTCAE v5.0 grade 1.
  * Exception: - clinically stable hypothyroid status managed with hormone replacement therapy, is permitted

Other Exclusions

* Female participant is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 6 months after the last dose of AMG 994 and/or AMG 404.
* Female participants of childbearing potential unwilling to use 1 highly effective method of contraception during treatment and for an additional 6 months after the last dose of AMG 994 and/or AMG 404.
* Female participants of childbearing potential with a positive pregnancy test assessed at day 1 by a serum pregnancy test.
* Male participants with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 8 months after the last dose of AMG 994 and/or AMG 404.
* Male participants unwilling to abstain from donating sperm during treatment and for an additional 8 months after the last dose of AMG 994 and/or AMG 404.
* Participant has known sensitivity to any of the products or components to be administered during dosing.
* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the participant and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to participant safety or interfere with the study evaluation, procedures or completion.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (17):
- United States (5):
  - City of Hope National Medical Center, Duarte, California
  - Henry Ford Hospital, Henry Ford Health Systems, Detroit, Michigan
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Monash Medical Centre, Clayton, Victoria
  - Linear Clinical Research Limited, Nedlands, Western Australia
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Centre Leon Berard, Lyon, France
- Germany (2):
  - Universitatsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
- Narodowy Instytut Onkologii im Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw, Poland
- Hospital Universitari Vall d Hebron, Barcelona, Catalonia, Spain
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 7 centers in Belgium, France, Japan, Poland, Spain, and the United States between 29 April 2021 and 05 June 2023.
Pre-assignment Details: The study was planned to be conducted in 2 parts: part 1 (dose exploration) and part 2 (dose expansion); however, no participants enrolled beyond Cohort 2 due to a business decision to discontinue development of AMG 994. This decision was unrelated to the safety or efficacy.
Groups:
- Cohort 1 (Low Dose): Participants were administered AMG 994 as a monotherapy treatment at dose level 1 (low dose) via short-term IV infusion once weekly (QW) for cycles 1 to 12 (on days 1, 8, 15, and 22). From Cycle 2, participants were also administered AMG 404 via short-term IV infusion every 4 weeks (Q4W) for up to 12 cycles (cycle= 28 days).
- Cohort 2 (High Dose): Participants were administered AMG 994 as a monotherapy treatment at dose level 2 (high dose) via short-term IV infusion QW for cycles 1 to 12 (on days 1, 8, 15, and 22). From Cycle 2, participants were also administered AMG 404 via short-term IV infusion Q4W for up to 12 cycles (cycle= 28 days).
Period: Overall Study
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Started | 3 | 8
Received AMG 994 | 3 | 8
Received AMG 404 | 3 | 6
Completed | 0 | 1
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 2 | 6
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: defined as all participants that are enrolled and receive at least 1 dose of AMG 994 or AMG 404.
Groups:
- Cohort 1 (Low Dose): Participants were administered AMG 994 as a monotherapy treatment at dose level 1 via short-term IV infusion QW for cycles 1 to 12 (on days 1, 8, 15, and 22). From Cycle 2, participants were also administered AMG 404 via short-term IV infusion Q4W for up to 12 cycles (cycle= 28 days).
- Cohort 2 (High Dose): Participants were administered AMG 994 as a monotherapy treatment at dose level 2 via short-term IV infusion QW for cycles 1 to 12 (on days 1, 8, 15, and 22). From Cycle 2, participants were also administered AMG 404 via short-term IV infusion Q4W for up to 12 cycles (cycle= 28 days).
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose) | Total
Number analyzed (Participants) | 3 | 8 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (7.2) | 61.1 (11.8) | 62.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 6 | 9
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 6 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs)
Description: DLTs were defined as:
  * Grade 5 events
  * Grade 4 neutropenia/thrombocytopenia of any duration
  * Grade 3 thrombocytopenia w/ clin significant bleeding or lasting >7 days
  * Febrile neutropenia
  * Grade 4 anemia
  * Grade 3/4 non-hematologic toxicity, except: Grade 3 nausea/vomiting or diarrhea < 72 hours; Grade 3 fatigue < 1 week; Asymptomatic grade 3 electrolyte abnormalities that last < 72 hours, are not clinically complicated, and resolve spontaneously or respond to conventional medical interventions; Grade 3 amylase/ lipase elevations; Other laboratory parameters of grade 3, not considered clinically relevant and improved to grade ≤ 2 within 72 hours.
  * Any grade 3 event requiring hospitalization
  * Recurrent grade 2 pneumonitis
  * Delay in cycle 2 treatment for > 14 days due to an adverse event in the dose escalation portion of the study
  * Any event requiring discontinuation of AMG 994
Time Frame: Up to Day 28 of Cycle 1 (one cycle = 28 days)
Population: Early DLT evaluable analysis set: included participants that were enrolled and received at least 1 dose of AMG 994 with an evaluable early DLT endpoint (evaluable in AMG 994 monotherapy cohort).
Measure: Number; unit: Number of participants
Groups:
- Cohort 2 (High Dose: Participants were administered AMG 994 as a monotherapy treatment at dose level 2 via short-term IV infusion QW for cycles 1 to 12 (on days 1, 8, 15, and 22). From Cycle 2, participants were also administered AMG 404 via short-term IV infusion Q4W for up to 12 cycles (cycle= 28 days).
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose
Number analyzed (Participants) | 3 | 8
Number of participants | 0 | 3

2. Primary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were those that occurred after the first intervention dose. A serious adverse event (SAE) included outcomes such as death, life-threatening situations, hospitalization or an extended hospital stay, significant incapacity, congenital defects, or other crucial medical events. AE severity followed the CTCAE Version 5.0 scale: grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (life-threatening), and grade 5 (death). Clinically significant laboratory results or other assessments (e.g., ECGs, scans, vital signs) that worsened from baseline and were deemed important by the investigator, independent of disease progression, were also considered.
Time Frame: From first dose of investigational product through 140 days after last dose (AMG 994 or AMG 404, whichever is later), or end of study (whichever is first); median (min, max) duration was 12.5 ( 1.48, 19.32) months.
Population: Safety analysis set: defined as all participants that are enrolled and receive at least 1 dose of AMG 994 or AMG 404.
Measure: Number; unit: Number of participants
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 8
Number of participants
  All TEAEs | 3 | 8
  All Grade ≥ 3 TEAEs | 3 | 6
  All SAEs | 3 | 6
  All Fatal AEs (FAEs) | 2 | 6
  All AMG 994 related TEAEs | 2 | 4
  AMG 994 related Grade ≥ 3 TEAEs | 0 | 1
  AMG 994 related SAEs | 0 | 0
  AMG 994 related FAEs | 0 | 0
  All AMG 404 related TEAEs | 1 | 4
  AMG 404 related TEAEs Grade ≥ 3 TEAEs | 0 | 1
  AMG 404 related SAEs | 0 | 0
  AMG 404 related FAEs | 0 | 0

3. Secondary Outcome: Objective Response (OR) Per Modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: OR was defined as achieving complete response (CR) or partial response (PR) per the modified RECIST 1.1 where CR is the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm and PR is at 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 19.32 months
Population: Safety analysis set: defined as all participants that are enrolled and receive at least 1 dose of AMG 994 or AMG 404.
Measure: Number; unit: Number of participants
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 8
Number of participants
  CR | 0 | 0
  PR | 0 | 2

4. Secondary Outcome: Duration of Response (DoR) Per Modified RECIST 1.1
Description: DoR was defined as the number of months between first OR to disease progression or death (due to any cause), whichever occurs first. Median and 95% CI estimates of survival time were based on the Kaplan-Meier analysis.
Time Frame: Up to approximately 19.32 months
Population: Safety analysis set: defined as all participants that are enrolled and receive at least 1 dose of AMG 994 or AMG 404. Only participants with response are included in duration of response analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 0 | 2
Months |  | 11.09 [11.05 to NA] — Upper limit not reached.

5. Secondary Outcome: Overall Survival (OS) Per Modified RECIST 1.1
Description: OS was defined as the time from initiation of AMG 994 until event of death due to any cause. Median and 95% CI estimates of survival time were based on the Kaplan-Meier analysis.
Time Frame: Up to approximately 19.32 months
Population: Safety analysis set: defined as all participants that are enrolled and receive at least 1 dose of AMG 994 or AMG 404.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 8
Months | 5.99 [5.03 to NA] — Upper CI limit not reached due to the low number of observations. | 12.50 [1.48 to NA] — Upper CI limit not reached due to the low number of observations.

6. Secondary Outcome: Progression-free Survival Per Modified RECIST 1.1
Description: PFS was defined as the time from initiation of AMG 994 until disease progression or death whichever occurs first. Death due to any cause counted as the event. Median and 95% CI estimates of survival time were based on the Kaplan-Meier analysis.
Time Frame: Up to approximately 19.32 months
Population: Safety analysis set: defined as all participants that are enrolled and receive at least 1 dose of AMG 994 or AMG 404.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 8
Months | 2.63 [2.63 to NA] — Upper CI limit not reached due to the low number of observations. | 1.61 [0.92 to 13.65]

7. Secondary Outcome: Time to Progression (TTP) Per Modified RECIST 1.1
Description: TTP was defined as time from initiation of AMG 994 until disease progression. Median and 95% CI estimates of survival time were based on the Kaplan-Meier analysis.
Time Frame: Up to approximately 19.32 months
Population: Safety analysis set: defined as all participants that are enrolled and receive at least 1 dose of AMG 994 or AMG 404.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 8
Months | 2.63 [2.63 to NA] — Upper CI limit not reached due to the low number of observations. | 1.74 [0.92 to 13.65]

8. Secondary Outcome: Time to Subsequent Therapy
Description: Time to subsequent therapy was defined as the time from initiation of AMG 994 until the first subsequent therapy. Median and 95% CI estimates of survival time were based on the Kaplan-Meier analysis.
Time Frame: Up to approximately 19.32 months
Population: Safety analysis set: defined as all participants that are enrolled and receive at least 1 dose of AMG 994 or AMG 404.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 8
Months | NA [4.74 to NA] — Median and upper CI limit not reached due to the low number of observations. | NA [16.64 to NA] — Median and upper CI limit not reached due to the low number of observations.

9. Secondary Outcome: Maximum Serum Concentration (Cmax) of AMG 994
Time Frame: Cycle 1 and 2, Day 1 (pre-dose, end of infusion [EOI], 2, 4.5, 6.5, and 12 hours post dose); Cycle 1, Day 22 (pre-dose, EOI, 6, and 12 hours post dose)
Population: Only participants with available data are included for each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 8
ng/mL
  Cycle 1, Day 1 | 667 (1150) | 2450 (1140)
  Cycle 1, Day 22: number analyzed (Participants) | 3 | 6
  Cycle 1, Day 22 | 4450 (3020) | 2550 (1290)
  Cycle 2, Day 1: number analyzed (Participants) | 3 | 5
  Cycle 2, Day 1 | 2340 (3180) | 2830 (1260)

10. Secondary Outcome: Time to Maximum Serum Concentration (Tmax) of AMG 994
Time Frame: as for outcome 9
Population: Only participants with available data are included for each time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 8
hours
  Cycle 1, Day 1 | 8.4 (15) | 1.4 (0.68)
  Cycle 1, Day 22: number analyzed (Participants) | 3 | 6
  Cycle 1, Day 22 | 3.7 (1.1) | 1.5 (0.74)
  Cycle 2, Day 1: number analyzed (Participants) | 3 | 5
  Cycle 2, Day 1 | 3.0 (0.0096) | 2.7 (2.0)

11. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of AMG 994
Time Frame: as for outcome 9
Population: Only participants with available data are included for each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 7
ng/mL
  Cycle 1, Day 1 | 0.00 (0.00) | 0.00 (0.00)
  Cycle 1, Day 22: number analyzed (Participants) | 3 | 6
  Cycle 1, Day 22 | 0.00 (0.00) | 0.00 (0.00)
  Cycle 2, Day 1: number analyzed (Participants) | 3 | 5
  Cycle 2, Day 1 | 0.00 (0.00) | 0.00 (0.00)

12. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast) of AMG 994
Time Frame: as for outcome 9
Population: Only participants with available data are included for each time point.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 8
h*ng/mL
  Cycle 1, Day 1: number analyzed (Participants) | 1 | 8
  Cycle 1, Day 1 | 12100 (NA) — SD not calculable when n=1 | 15000 (16700)
  Cycle 1, Day 22: number analyzed (Participants) | 3 | 6
  Cycle 1, Day 22 | 18900 (15000) | 21900 (23100)
  Cycle 2, Day 1: number analyzed (Participants) | 3 | 5
  Cycle 2, Day 1 | 6460 (8010) | 22900 (23300)

13. Secondary Outcome: Area Under the Serum Concentration-time Curve During a Dosing Interval (AUCtau) of AMG 994
Time Frame: as for outcome 9
Population: Only participants with available data are included for each time point.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 7
h*ng/mL
  Cycle 1, Day 1 | 20300 (35200) | 20400 (21400)
  Cycle 1, Day 22: number analyzed (Participants) | 3 | 5
  Cycle 1, Day 22 | 24500 (18400) | 45400 (61100)
  Cycle 2, Day 1: number analyzed (Participants) | 3 | 5
  Cycle 2, Day 1 | 8260 (10100) | 29500 (31100)

14. Secondary Outcome: Terminal Half-life (t1/2) of AMG 994
Time Frame: as for outcome 9
Population: Only participants with available data are included for each time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 1 | 3
hours
  Cycle 1, Day 1: number analyzed (Participants) | 0 | 3
  Cycle 1, Day 1 |  | 4.97 (2.90)
  Cycle 1, Day 22: number analyzed (Participants) | 1 | 0
  Cycle 1, Day 22 | 5.24 (NA) — SD not calculable when n=1 |
  Cycle 2, Day 1: number analyzed (Participants) | 0 | 3
  Cycle 2, Day 1 |  | 4.76 (3.55)

15. Secondary Outcome: Cmax of AMG 404
Time Frame: Cycle 2, Day 1 (pre-dose, end of infusion [EOI], 2, 4.5, 6.5, and 12 hours post dose)
Population: Only participants with available data are included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 5
ng/mL | 158 (22.1) | 145 (47.9)

16. Secondary Outcome: Tmax of AMG 404
Time Frame: Cycle 2, Day 1 (pre-dose, end of infusion [EOI], 2, 4.5, 6.5, and 12 hours post dose)
Population: Only participants with available data are included.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 5
hours | 0.080 (0.049) | 0.11 (0.074)

17. Secondary Outcome: Cmin of AMG 404
Time Frame: Cycle 2, Day 1 (pre-dose, end of infusion [EOI], 2, 4.5, 6.5, and 12 hours post dose)
Population: Only participants with available data are included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 3
ng/mL | 20.8 (11.1) | 22.8 (18.2)

18. Secondary Outcome: AUClast of AMG 404
Time Frame: Cycle 2, Day 1 (pre-dose, end of infusion [EOI], 2, 4.5, 6.5, and 12 hours post dose)
Population: Only participants with available data are included.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 5
h*ng/mL | 1280 (322) | 1160 (618)

19. Secondary Outcome: AUCtau of AMG 404
Time Frame: Cycle 2, Day 1 (pre-dose, end of infusion [EOI], 2, 4.5, 6.5, and 12 hours post dose)
Population: Only participants with available data are included.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 3 | 5
h*ng/mL | 1280 (322) | 1290 (576)

20. Secondary Outcome: T1/2 of AMG 404
Time Frame: Cycle 2, Day 1 (pre-dose, end of infusion [EOI], 2, 4.5, 6.5, and 12 hours post dose)
Population: Only participants with available data are included.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
Number analyzed (Participants) | 1 | 1
hours | 13.0 (NA) — SD not calculable when n=1 | 9.55 (NA) — SD not calculable when n=1

ADVERSE EVENTS:
Time Frame: Serious and other AEs were collected from first dose of investigational product (IP) through 140 days after last dose of IP (AMG 994 or AMG 404, whichever is later), or end of study (whichever is first); median (min, max) duration was 12.5 ( 1.48, 19.32) months. ACM= from enrollment through end of study; median (min, max) time on study was 5.8 (1.48, 19.32) months.
Description: All-Cause Mortality was collected for all participants enrolled. Serious and other (Not Including Serious Adverse Events) were collected for all participants that received at least one dose of IP.
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (High Dose)
All-Cause Mortality (participants affected / at risk) | 2/3 | 6/8
Serious Adverse Events (participants affected / at risk) | 3/3 | 6/8
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Low Dose) (N=3) | Cohort 2 (High Dose) (N=8)
Coronary artery disease (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Epithelioid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Low Dose) (N=3) | Cohort 2 (High Dose) (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 1
Rectal fissure (Gastrointestinal disorders) | 0 | 1
Tongue geographic (Gastrointestinal disorders) | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 0 | 2
Axillary pain (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 2
Fatigue (General disorders) | 2 | 2
Impaired healing (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Hepatic pain (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Retinitis viral (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatine increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Peripheral coldness (Vascular disorders) | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was planned to be conducted in 2 parts: part 1 (dose exploration) and part 2 (dose expansion); however, no participants enrolled beyond Cohort 2 due to a business decision to discontinue development of AMG 994. This decision was unrelated to the safety or efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT04727554/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT04727554/SAP_001.pdf